CLINICAL TRIAL: NCT03001973
Title: High Quality Evidence of Chinese Lupus Nephritis (HELP)
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xue Qing Yu, Professor, Sun Yat-sen University
Other Study IDs: HELP
Record Dates: First submitted 2016-12-21; First posted 2016-12-23 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Lupus Nephritis
Keywords: Lupus nephritis; Patient survival; Renal survival
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The serum, urine, DNA and renal tissue will be collected.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- LN patients: Patients diagnosis as lupus nephritis
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — Registration of all LN patients in the First Affiliated Hospital of Sun Yat-sen University and other hospitals which have signed the contract in China.

SUMMARY:
The investigators are registering LN patients at recruited hospitals and developing a LN database in China. Patients will be follow-up every year, and both baseline and follow-up information will be entered into the registration system.

DETAILED DESCRIPTION:
The investigators are registering Lupus nephritis (LN) and developing a LN database in China. Patients' demographic characteristics (including age, gender, height, weight, BMI, smoking, drinking, and education etc.), clinical characteristics (including systolic blood pressure, diastolic blood pressure, and lab measurements of whole blood, serum, urine etc.), complications, drug information at the baseline will be collected. Patients will be follow-up every year, the demographic and clinical characteristics, complications; drug information of patients will be collected at each visit. We will also record the outcome at each visit, such as mortality (including all-cause mortality and cardiovascular disease mortality), end-stage renal disease (ESRD) or serum creatinine doubling. The patient survival and renal survival will be compared using the LN database.

ELIGIBILITY:
Inclusion Criteria:

* Patients who diagnosis as lupus nephritis

Exclusion Criteria:

* No

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Lupus nephritis patients
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2013-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality and cardiovascular mortality of LN patients | 10years
A composite renal outcome of LN patients | 10years
  The composite renal outcome defined as doubling of serum creatinine and ESRD (defined as initiation of dialysis or kidney transplantation).

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Tian N, Zhou Q, Yin P, Chen W, Hong L, Luo Q, Chen M, Yu X, Chen W. Long-Term Kidney Prognosis and Pathological Characteristics of Late-Onset Lupus Nephritis. Front Med (Lausanne). 2022 May 30;9:882692. doi: 10.3389/fmed.2022.882692. eCollection 2022. PMID 35712095
- [Derived] Yin P, Zhou Y, Li B, Hong L, Chen W, Yu X. Effect of low and high HDL-C levels on the prognosis of lupus nephritis patients: a prospective cohort study. Lipids Health Dis. 2017 Dec 6;16(1):232. doi: 10.1186/s12944-017-0622-3. PMID 29212518